CLINICAL TRIAL: NCT00978068
Title: A Randomized Open Label Trial of HIV Protease Inhibitors for the Prevention of Malaria in HIV-Infected Children
Brief Title: HIV Protease Inhibitors for the Prevention of Malaria in Ugandan Children
Acronym: PROMOTE-PEDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H5747-34097; NIH PO1 HD059454; 2009-114 (Other: Makerere Univ Fac of Med Research and Ethics Committee); HS-620 (Other: Uganda National Council for Science and Tech); 551/ESR/NDA/DID-08/09 (Other: Uganda National Drug Authority); H5741-34097 and 10-00991 (Other: UCSF Committee on Human Research)
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Malaria; HIV Infections
Keywords: Pediatric HIV; Malaria; Uganda; Nevirapine; Zidovudine; Lamivudine; Lopinavir/ritonavir; Stavudine; Efavirenz; HIV
MeSH Terms: conditions — Malaria; HIV Infections | interventions — Lopinavir; lopinavir-ritonavir drug combination; Nevirapine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lopinavir/ritonavir (LPV/r) +2 NRTI (Active Comparator): Lopinavir/ritonavir (LPV/r) +2 nucleoside reverse transcriptase inhibitor (NRTI)
  Interventions: Drug: Lopinavir/Ritonavir (LPV/r); Drug: 2 nucleoside reverse transcriptase inhibitor (NRTI)
- Nevirapine (NVP) or Efavirenz (EFV) +2 NRTI (Active Comparator): Nevirapine (NVP) or Efavirenz (EFV) +2 nucleoside reverse transcriptase inhibitor (NRTI)
  Interventions: Drug: Nevirapine (NVP); Drug: Efavirenz (EFV); Drug: 2 nucleoside reverse transcriptase inhibitor (NRTI)

INTERVENTIONS:
Drug: Lopinavir/Ritonavir (LPV/r)
  Other Names: Aluvia
  Arms: Lopinavir/ritonavir (LPV/r) +2 NRTI
Drug: Nevirapine (NVP) — NVP will be used for children < 3 years of age
  Arms: Nevirapine (NVP) or Efavirenz (EFV) +2 NRTI
Drug: Efavirenz (EFV) — EFV for children ≥3 years of age
  Arms: Nevirapine (NVP) or Efavirenz (EFV) +2 NRTI
Drug: 2 nucleoside reverse transcriptase inhibitor (NRTI) — The same NRTI choice strategy will be used for both arms. Lamivudine will be used with all children. The second NRTI will be zidovudine unless the participant has a hemoglobin < 8 gm/dL, in which case it will be Abacavir. Stavudine will be used in the event that a participant is unable to take Abacavir for safety or other reasons.

SUMMARY:
HIV and malaria are major causes of morbidity and mortality in Sub-Saharan Africa and children bear the greatest brunt of both diseases. No single existing intervention is likely to control malaria in Africa. Rather, improvements in malaria prevention are likely to come from strategies that employ multiple proven interventions targeting different populations. HIV-infected children represent one of the most vulnerable subpopulations in these countries. It is possible that the use of protease inhibitor (PI) - based antiretroviral therapy (ART) in HIV-infected children living in areas of high malaria transmission could prevent malaria in this vulnerable population. An effective remedy that offers the possibility to further reduce malaria risk, such as PIs, is highly desirable. This study will determine whether a PI based ART regimen will reduce malaria among children living in a malaria endemic area of Uganda and receiving insecticide-treated bed nets (ITN) and TS. This study will compare two different ART regimens. Children enrolled in the study will start or continue to receive either standard Ugandan first line treatment ART regimen (NNRTI+2 NRTIs) or an ART regimen containing the HIV protease inhibitor (lopinavir/ritonavir +2 NRTIs) and followed for a period of 24 months.

DETAILED DESCRIPTION:
This is an open label, single site, randomized clinical trial comparing PI-based ART to NNRTI-based ART for the prevention of malaria in HIV-infected children. The two ART drug regimens that will be used include: Treatment arm 1. LPV/r + 2 NRTIs and Treatment arm 2. NVP or EFV + 2 NRTIs. The study is designed to test the hypothesis that children receiving a PI-based ART regimen will have lower the incidence of malaria compared to children receiving an NNRTI- based ART regimen. The primary study endpoint of the study is malaria incidence.

The study site will be the Tororo District Hospital campus situated in Eastern Uganda, an area of high malaria transmission. Using convenience sampling, 300 HIV-infected children identified from the Tororo community aged 2 months to <11 years either eligible for ART-initiation or already receiving a first line ART regimen with HIV RNA<400 copies/ml will be evaluated for enrollment.

Eligible children will be randomized at enrollment to receive either a PI- based or an NNRTI-based ART regimen. At enrollment, all study participants will receive a long lasting ITN as part of a basic care package including a safe water vessel and multivitamins and given TS chemoprophylaxis, as per current standard of care for HIV-infected children in Uganda. On the day of ART initiation, patients will be counseled about the importance of adherence to ART and possible ART related toxicities. After 2 weeks, patients will be seen to assess adherence and toxicity to study medications by interview and clinical examination. Apart from this visit at week 2, patients will be seen at 4 week intervals timed from ART-initiation. Assessment of adherence will also be done for TS prophylaxis, ITN use and ART. Assessment of adherence to ART will be done by self report of missed doses and pill counts.

Participants will receive all routine and acute medical care at a designated study clinic open 7 days a week from 8 a.m. to 5 p.m. Parents/guardians will be asked to bring their child to the study clinic for all medical care. If after hours, they will be instructed to bring them to Tororo District Hospital premises (where the study clinic is located) and request that the study physician on-call be contacted. They will be followed for at least 24 months and up to 3 years. They will be seen monthly for routine assessments with laboratory evaluations done at every 3 months. At these visits, the study protocol will be reinforced with discussion regarding the need to come to the study clinic promptly upon the onset of any illness and to avoid use of outside medications. Study participants will also be followed closely for adverse events potentially due to study drugs and for malaria and HIV treatment outcomes. During the follow-up period, all patients presenting to the clinic with a new episode of fever will undergo standard evaluation (history, physical examination) and Giemsa-stained blood smear for the diagnosis of malaria.

ELIGIBILITY:
Inclusion criteria:

1. Age 2 months to < 11 years
2. Confirmed HIV diagnosis. i. Children > 18 months: Documentation of HIV status must come from two assays. Assays include DNA PCR, HIV RNA, Western blot, or rapid HIV antibody test ii. Children < 18 months: Documentation will be DNA PCR confirmation only along with documentation of testing from the referral entity
3. ART-naïve patients eligible for ART initiation per WHO/Uganda guidelines (see Table 1) or Patients receiving first line ART regimen with NNRTI +2 NRTI with at least one HIV RNA <400 copies/ml within the past 6 months
4. Agreement to come to the study clinic for any febrile episode or other illness
5. Agreement to avoid medications administered outside study protocol
6. Provision of informed consent by parent/guardian and agreement to have child's care at the clinical site
7. Lives within 50 km of study site

Exclusion criteria:

1. ART-naïve children: children or their mothers that have received any dose of Nevirapine in the past 24 months
2. Active medical problem requiring in-patient evaluation at the time of screening or enrollment
3. History of cardiac conduction disorder or known significant cardiac structural defect
4. Children receiving any disallowed medications (see section 4.3)
5. Moderate, Severe or Life-threatening (Grade 2, 3, or 4) AST or ALT found within 4 weeks prior to enrollment:

   * AST: >113U/L (>2.5xULN)
   * ALT: >113U/L (>2.5xULN)
6. Life-threatening (Grade 4) screening laboratory value found within 4 weeks prior to enrollment for the following:

   * Absolute neutrophil count: <500 mm3
   * Hemoglobin: <6.5 g/dL
   * Creatinine: >3.5xULN
   * Platelets: <25,000/mm3

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane V Havlir, MD, Study Director — University of California, San Francisco; Moses R Kamya MBChB, MMed, MPH, Principal Investigator — Makerere University; Grant Dorsey, MD, PhD, Principal Investigator — University of California, San Francisco; Ted Ruel, MD, Principal Investigator — University of California, San Francisco; Jane Achan, MBChB, MPed, Principal Investigator — Makerere University
Locations (1):
- IDRC - Tororo Research Clinic, Tororo, Uganda

REFERENCES:
- [Result] Achan J, Kakuru A, Ikilezi G, Ruel T, Clark TD, Nsanzabana C, Charlebois E, Aweeka F, Dorsey G, Rosenthal PJ, Havlir D, Kamya MR. Antiretroviral agents and prevention of malaria in HIV-infected Ugandan children. N Engl J Med. 2012 Nov 29;367(22):2110-8. doi: 10.1056/NEJMoa1200501. PMID 23190222
- [Result] Ikilezi G, Achan J, Kakuru A, Ruel T, Charlebois E, Clark TD, Rosenthal PJ, Havlir D, Kamya MR, Dorsey G. Prevalence of asymptomatic parasitemia and gametocytemia among HIV-infected Ugandan children randomized to receive different antiretroviral therapies. Am J Trop Med Hyg. 2013 Apr;88(4):744-6. doi: 10.4269/ajtmh.12-0658. Epub 2013 Jan 28. PMID 23358639
- [Result] Nsanzabana C, Rosenthal PJ. In vitro activity of antiretroviral drugs against Plasmodium falciparum. Antimicrob Agents Chemother. 2011 Nov;55(11):5073-7. doi: 10.1128/AAC.05130-11. Epub 2011 Aug 29. PMID 21876053
- [Result] Ruel TD, Kakuru A, Ikilezi G, Mwangwa F, Dorsey G, Rosenthal PJ, Charlebois E, Havlir D, Kamya M, Achan J. Virologic and immunologic outcomes of HIV-infected Ugandan children randomized to lopinavir/ritonavir or nonnucleoside reverse transcriptase inhibitor therapy. J Acquir Immune Defic Syndr. 2014 Apr 15;65(5):535-41. doi: 10.1097/QAI.0000000000000071. PMID 24326597
- [Result] Kakuru A, Achan J, Muhindo MK, Ikilezi G, Arinaitwe E, Mwangwa F, Ruel T, Clark TD, Charlebois E, Rosenthal PJ, Havlir D, Kamya MR, Tappero JW, Dorsey G. Artemisinin-based combination therapies are efficacious and safe for treatment of uncomplicated malaria in HIV-infected Ugandan children. Clin Infect Dis. 2014 Aug 1;59(3):446-53. doi: 10.1093/cid/ciu286. Epub 2014 Apr 23. PMID 24759826
- [Result] Bartelink IH, Savic RM, Dorsey G, Ruel T, Gingrich D, Scherpbier HJ, Capparelli E, Jullien V, Young SL, Achan J, Plenty A, Charlebois E, Kamya M, Havlir D, Aweeka F. The effect of malnutrition on the pharmacokinetics and virologic outcomes of lopinavir, efavirenz and nevirapine in food insecure HIV-infected children in Tororo, Uganda. Pediatr Infect Dis J. 2015 Mar;34(3):e63-70. doi: 10.1097/INF.0000000000000603. PMID 25742090
- [Result] Achan J, Kakuru A, Ikilezi G, Mwangwa F, Plenty A, Charlebois E, Young S, Havlir D, Kamya M, Ruel T. Growth Recovery Among HIV-infected Children Randomized to Lopinavir/Ritonavir or NNRTI-based Antiretroviral Therapy. Pediatr Infect Dis J. 2016 Dec;35(12):1329-1332. doi: 10.1097/INF.0000000000001318. PMID 27580060
- [Derived] Bangirana P, Ruel TD, Boivin MJ, Pillai SK, Giron LB, Sikorskii A, Banik A, Achan J. Absence of neurocognitive disadvantage associated with paediatric HIV subtype A infection in children on antiretroviral therapy. J Int AIDS Soc. 2017 Oct;20(2):e25015. doi: 10.1002/jia2.25015. PMID 29052340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from September 2009 through July 2011.
Pre-assignment Details: A total of 404 children were screened for eligibility; 228 were found not to be eligible. The main reasons for ineligibility were:
  136 Were not eligible for ART 34 Were on ART with detectable viral load 32 Were HIV- 8 Had not received ART but had prior exposure to nevirapine
Groups:
- LPV/r + 2 NRTIs: LPV/r + 2 NRTIs: Group 1
  Lopinavir/ritonavir (LPV/r) +2 nucleoside reverse transcriptase inhibitor (NRTI)
  The same NRTI choice strategy will be used for both arms. Lamivudine will be used with all children. The second NRTI will be zidovudine unless the participant has a hemoglobin < 8 gm/dL, in which case it will be Abacavir. Stavudine will be used in the event that a participant is unable to take Abacavir for safety or other reasons.
- NVP or EFV + 2 NRTIs: NVP or EFV + 2 NRTIs: Group 2
  Nevirapine (NVP) or Efavirenz (EFV) + 2 NRTI
  NVP will be used for children < 3 years of age and EFV for children ≥3 years of age. The same NRTI choice strategy will be used for both arms. Lamivudine will be used with all children. The second NRTI will be zidovudine unless the participant has a hemoglobin < 8 gm/dL, in which case it will be stavudine.
Period: Overall Study
Arm/Group | LPV/r + 2 NRTIs | NVP or EFV + 2 NRTIs
Started | 87 | 89
Initiated Study Drugs | 84 | 86
Completed | 83 | 80
Not Completed | 4 | 9
Not completed — Were Awaiting Initiation of ART | 2 | 2
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Unable to Comply with Study | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LPV/r + 2 NRTIs | NVP or EFV + 2 NRTIs | Total
Number analyzed (Participants) | 84 | 86 | 170
Age, Continuous [Median (Full Range); unit: years] | 2.9 [0.7 to 6.0] | 3.1 [0.5 to 5.9] | 3.1 [0.5 to 6.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 82
  Male | 43 | 45 | 88
Previous ART to Enrollment [Number; unit: participants]
  No Previous ART | 57 | 58 | 115
  Previous ART | 27 | 28 | 55
WHO Clinical HIV stage [Number; unit: participants] — clinical staging is based on standard WHO grading scales found is the document: https://www.who.int/hiv/pub/guidelines/clinicalstaging.pdf
  participants
    Stage I (Asymptomatic) | 60 | 66 | 126
    Stage II (mod. unexplained weight loss) | 16 | 15 | 31
    Stage III (unexplained severe weight loss) | 2 | 1 | 3
    Stage IV (HIV wasting syndrome) | 6 | 4 | 10
CD4 Percentage [Median (Full Range); unit: % of white cells that are CD4 cells] — The percentage represents the percentage of white cells that are CD4 cells.
  % of white cells that are CD4 cells
    No Previous ART | 14 [2 to 44] | 16 [2 to 43] | 16 [2 to 44]
    Previous ART | 31 [8 to 51] | 30 [10 to 45] | 30 [8 to 51]
Viral Load [Median (Full Range); unit: log10copies/mL] — 0 = below the level of detection (<400 copies per microliter).
  log10copies/mL
    No Previous ART | 5.4 [0 to 6.4] | 5.5 [0 to 6.4] | 5.5 [0 to 6.4]
    Previous ART | NA [NA to NA] — Below the level of detection (<400 copies per microliter) | NA [NA to NA] — Below the level of detection (<400 copies per microliter) | NA [NA to NA] — Below the level of detection (<400 copies per microliter)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 10.4 (1.3) | 10.6 (1.5) | 10.5 (1.4)
Result of Baseline Blood Smear for Asexual Parasites [Number; unit: participants]
  Positive | 10 | 11 | 21
  Negative | 74 | 75 | 149

OUTCOME MEASURES:

1. Primary Outcome: Incidence-density of Malaria Defined as the Number of Incident Episodes of Malaria Per Time at Risk.
Time Frame: Time from randomization to at least 24 months of follow up or until end of the study
Measure: Number; unit: Episodes/ Person-Yr at Risk
Groups:
- Group 1: LPV/r + 2 NRTIs: Lopinavir/ritonavir (LPV/r) +2 nucleoside reverse transcriptase inhibitor (NRTI)
  The same NRTI choice strategy will be used for both arms. Lamivudine will be used with all children. The second NRTI will be zidovudine unless the participant has a hemoglobin < 8 gm/dL, in which case it will be Abacavir. Stavudine will be used in the event that a participant is unable to take Abacavir for safety or other reasons.
- Group 2: Nevirapine (NVP) or Efavirenz (EFV) + 2 NRTIs: NVP will be used for children < 3 years of age and EFV for children ≥3 years of age. The same NRTI choice strategy will be used for both arms. Lamivudine will be used with all children. The second NRTI will be zidovudine unless the participant has a hemoglobin < 8 gm/dL, in which case it will be stavudine.
Arm/Group | Group 1: LPV/r + 2 NRTIs | Group 2: Nevirapine (NVP) or Efavirenz (EFV) + 2 NRTIs
Number analyzed (Participants) | 84 | 86
Episodes/ Person-Yr at Risk | 1.32 | 2.25
Statistical Analysis 1: Comparison: Group 1: LPV/r + 2 NRTIs vs Group 2: Nevirapine (NVP) or Efavirenz (EFV) + 2 NRTIs; We assumed that the incidence of malaria in Group 2 would be 0.70 episodes per person-year and estimated that we would need a sample of 300 participants for the study to have 80% power to show a 35% reduction in the incidence of malaria in Group 1, at a 2-sided significance level of 0.05. We then observed an incidence of malaria in Group 2 that was higher than anticipated (2.19 episodes/person-yr) and revised the sample size to 150 participants, who would be followed for at least 6 months; Test type: Superiority or Other; p = 0.04, Negative Binomial Regression; Incidence Rate Ratio = 0.59, 95% CI 2-sided [0.36 to 0.97] — Group 1 represents the numerator for the rate ratio. Group 2 represents the denominator for the rate ratio

2. Secondary Outcome: Percentage of Uncomplicated Malaria Episodes With Accompanying Adverse Events That Occurred in the 28 Days Following Antimalarial Therapy
Description: The rates of adverse events, defined as severity grade 2 or higher that are possibly, probably or definitely related to study drugs over the course of the 28-day period after antimalarial therapy with artemether-lumefantrine (AL).
Time Frame: 28 days after antimalarial therapy
Measure: Number; unit: % uncomplicated malaria episodes w/ AEs
Arm/Group | LPV/r + 2 NRTIs | NVP or EFV + 2 NRTIs
Number analyzed (Participants) | 84 | 86
% uncomplicated malaria episodes w/ AEs | 71.0 | 79.3
Statistical Analysis 1: Comparison: LPV/r + 2 NRTIs vs NVP or EFV + 2 NRTIs; Test type: Superiority or Other; p = 0.13, Cox Proportional-Hazards

3. Secondary Outcome: Incidence-density of Malaria Defined as the Number of Incident Episodes of Complicated Malaria Per Time at Risk.
Time Frame: Time from randomization to at least 24 months of follow up or until end of the study
Measure: Number; unit: Episodes/ Person-Yr at Risk
Groups:
- Group 1: LPV/r + 2 NRTIs
  LPV/r + 2 NRTIs: Group 1
  Lopinavir/ritonavir (LPV/r) +2 nucleoside reverse transcriptase inhibitor (NRTI)
  The same NRTI choice strategy will be used for both arms. Lamivudine will be used with all children. The second NRTI will be zidovudine unless the participant has a hemoglobin < 8 gm/dL, in which case it will be Abacavir. Stavudine will be used in the event that a participant is unable to take Abacavir for safety or other reasons.
- Group 2: NVP or EFV + 2 NRTIs
  NVP or EFV + 2 NRTIs: Group 2
  Nevirapine (NVP) or Efavirenz (EFV) + 2 NRTI
  NVP will be used for children < 3 years of age and EFV for children ≥3 years of age. The same NRTI choice strategy will be used for both arms. Lamivudine will be used with all children. The second NRTI will be zidovudine unless the participant has a hemoglobin < 8 gm/dL, in which case it will be stavudine.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 84 | 86
Episodes/ Person-Yr at Risk | 0.024 | 0.026
Statistical Analysis 1: Comparison: Group 1 vs Group 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.87, Negative Binomial Regression; Incidence Rate Ratio = 0.80, 95% CI 2-sided [0.06 to 11.16] — Group 1 represents the numerator for the rate ratio. Group 2 represents the denominator for the rate ratio

4. Secondary Outcome: Estimates of the 6-month Risk of a First Episode of Malaria
Description: To assess the effect of ART independently of potential interactions with antimalarial therapy after treatment for malaria, we compared the two groups with respect to the time to the first episode of malaria. Cumulative risk was estimated using the Kaplan-Meier product-limit formula.
Time Frame: Enrollment to 6 months follow up
Population: Among patients who were followed for 6 months, malaria did not develop in 34 patients in the NNRTI group and 44 in the lopinavir-ritonavir group; data on 10 patients in the NNRTI group and 7 in the lopinavir-ritonavir group were censored before the 6-month follow-up assessment.
Measure: Number (95% Confidence Interval); unit: Cumulative Risk Percentage
Arm/Group | LPV/r + 2 NRTIs | NVP or EFV + 2 NRTIs
Number analyzed (Participants) | 84 | 86
Cumulative Risk Percentage | 40.7 [30.9 to 52.2] | 52.5 [42.0 to 63.9]
Statistical Analysis 1: Comparison: LPV/r + 2 NRTIs vs NVP or EFV + 2 NRTIs; Test type: Superiority or Other; p = 0.14, Cox Proportional-Hazards; Adjustment for repeated measures in the same patient; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.45 to 1.12] — Group 1 represents the numerator for the hazard ratio. Group 2 represents the denominator for the hazard ratio

5. Secondary Outcome: 28-day Risk of Recurrent Parasitemia
Description: To assess the effect of potential interactions between ART and artemether-lumefantrine, the risks of recurrent parasitemia at 28 days were compared between the two groups.
Time Frame: 28 days after antimalarial therapy
Population: The risk of recurrence was assessed among patients who had had uncomplicated malaria that had been treated with artemether-lumefantrine.
Measure: Number (95% Confidence Interval); unit: Cummulative Risk Percentage
Arm/Group | LPV/r + 2 NRTIs | NVP or EFV + 2 NRTIs
Number analyzed (Participants) | 84 | 86
Cummulative Risk Percentage | 14.0 [8.7 to 22.2] | 40.8 [33.9 to 48.6]
Statistical Analysis 1: Comparison: LPV/r + 2 NRTIs vs NVP or EFV + 2 NRTIs; Test type: Superiority or Other; p = 0.004, Cox Proportional-Hazards; Adjustment for repeated measures in same participant; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.14 to 0.68] — Group 1 represents the numerator for the hazard ratio. Group 2 represents the denominator for the hazard ratio

6. Secondary Outcome: 63-day Risk of Recurrent Malaria
Description: To assess the effect of potential interactions between ART and artemether-lumefantrine, the risks of recurrent malaria at 63 days were compared between the two groups.
Time Frame: 28 days after antimalarial therapy
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Cumulative Risk Percentage
Arm/Group | LPV/r + 2 NRTIs | NVP or EFV + 2 NRTIs
Number analyzed (Participants) | 84 | 86
Cumulative Risk Percentage | 28.1 [20.2 to 38.3] | 54.2 [46.4 to 62.2]
Statistical Analysis 1: Comparison: LPV/r + 2 NRTIs vs NVP or EFV + 2 NRTIs; Test type: Superiority or Other; p = 0.004, Cox Proportional-Hazards; Adjustment for repeated measures in the same patient; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.22 to 0.76] — Group 1 represents the numerator in the hazard ratio. Group 2 represents the denominator in the hazard ratio

ADVERSE EVENTS:
Time Frame: Time from randomization to at least 24 months of follow up or until end of the study
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 11/84 | 9/86
Other Adverse Events (participants affected / at risk) | 41/84 | 43/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=84) | Group 2 (N=86)
Anemia (Blood and lymphatic system disorders) | 2 | 3
Altered mental status (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dehydration (Blood and lymphatic system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dyspnea/respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Elevated ALT (Hepatobiliary disorders) | 2 | 2
Elevated Temperature/Fever (Endocrine disorders) | 2 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Neutropenia/Absolute neutrophil count (Blood and lymphatic system disorders) | 7 | 9
Seizure (Nervous system disorders) | 2 | 1
Hypoglycemia (Renal and urinary disorders) | 0 | 1
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombocytopenia Platelets, decreased (Blood and lymphatic system disorders) | 3 | 1
Unintentional weight loss (Metabolism and nutrition disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=84) | Group 2 (N=86)
Anemia (Blood and lymphatic system disorders) | 2 | 4
Chills (Endocrine disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Elevated ALT (Hepatobiliary disorders) | 2 | 3
Elevated AST (Hepatobiliary disorders) | 1 | 1
Elevated Temperature (Endocrine disorders) | 19 | 24
Neutropenia (Blood and lymphatic system disorders) | 24 | 21
Pallor (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (non-infectious) (Skin and subcutaneous tissue disorders) | 0 | 1
Severe Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Thrombocytopenia Platelets, decreased (Blood and lymphatic system disorders) | 9 | 6
Unintentional weight loss (Metabolism and nutrition disorders) | 1 | 0
WBC, decreased (Blood and lymphatic system disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
The study has limited statistical power for the comparison of uncommon events and limited evaluation of potential cardiotoxic effects, hence future studies of the safety of coadministration of lopinavir-ritonavir and lumefantrine are warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No